CLINICAL TRIAL: NCT03579589
Title: The Effect of Sugammadex Versus Neostigmine During Neuromuscular Blockade Reversal in Outpatient Surgeries - An Evaluation of Clinical and Associated Health Care Cost
Brief Title: The Effect of Sugammadex Versus Neostigmine During Neuromuscular Blockade Reversal
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Jarrett Heard, M.D., Principal INvestigator, Clinical Assitant Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018H0102
Record Dates: First submitted 2018-04-03; First posted 2018-07-06 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Neuromuscular Blockade
Keywords: Neuromuscular Blockade Reversal; Outpatient Surgery

STUDY DESIGN:
Intervention Model Description: Sugammadex vs Neostigmine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sugammadex (Active Comparator): * If spontaneous recovery has reached second twitch after TOF: 2 mg/kg
  * If spontaneous recovery has reached between 1-2 post-tetanic counts but no twitch responses to TOF: 4 mg/kg
  * When there is a clinical need to reverse NMB within 3 min of a single dose of rocuronium (1.2 mg/kg): 16 mg/kg
  Interventions: Drug: Sugammadex vs Neostigmine
- Neostigmine (Active Comparator): 50 µg. Kg-1 will be administered after spontaneous recovery has reached fourth twitch after TOF in accordance with our institutional standard procedures and published literature.
  Interventions: Drug: Sugammadex vs Neostigmine

INTERVENTIONS:
Drug: Sugammadex vs Neostigmine — Patients will be randomized into either Sugammadex or Neostigmine neuromuscular blockade reversal.

SUMMARY:
Patients who undergo surgery receive drugs called neuromuscular blocking agents (NMBA) that to block the activity of muscles. When the surgery is over, the block needs to be reversed. Suggammadex and neostigmine are examples of drugs that reverse blocks. This study aims to investigate if sugammadex is associated with a significantly reduced time to discharge from the operating room to the postoperative unit when compared to neostigmine.

DETAILED DESCRIPTION:
This is a single-center, randomized, double arm prospective clinical trial involving adult patients undergoing outpatient surgeries at The OSUWMC. Institutional review board (Office of Responsible Research practices) approval is mandatory preceding the start of the clinical trial. Written informed consent will be obtained from all eligible patients participating in this trial, and signed prior to the initiation of any study-related procedures. The study will be conducted in accordance with the principles of Good Clinical Practice and will be approved by the appropriate institutional review boards at OSUWMC. An individual with appropriate human subjects protection and HIPAA education will undertake the consent process in the surgeon's office or other appropriate location (e.g. preoperative clinics). Researchers will utilize the electronic medical record (EMR) to screen and identify surgical cases based on study inclusion criteria. These cases will be reviewed together with the surgical team to determine whether all inclusion and exclusion criteria are met, prior to approaching the patient. Prior surgery, a study-team investigator will approach the patient to discuss the nature of the study, its requirements, and potential risks. Written informed consent will be obtained from every subject prior to the start any study related procedures and enough time will be allowed for the subject to ask questions and receive answers. The inclusion and exclusion criteria will be reviewed in order to ascertain whether a patient qualifies for this study. Subjects must meet all the inclusion criteria and none of the exclusion criteria to qualify for the study.

* All medication taken 7 days prior surgery will be recorded. Demographic information, previous medical history, vital signs, urine pregnancy test, and a physical examination will be performed at this time as a standard of care and results will be recorded.
* Study medication dosages will be calculated prior to surgery by using total body weight (TBW) by the research team, following standard operational procedures.

II.4.B. Intraoperative phase

* Pre-induction: intravenous midazolam (2 - 4 mg) if required.
* Induction of general anesthesia: anesthesia will follow the standard of care protocols set by our center. Therefore, preoxygenation will be achieved with 100% oxygenation for at least 5 full Tidal Volume and suggested dosage of anesthetic drugs will be as follows: propofol 1-2 mg/kg, lidocaine IV 40-100 mg, fentanyl IV 1-2 μg/Kg, and sevoflurane 0.5-1 MAC (if needed). Additionally, rocuronium (0.3-0.7 mg/kg) will be used for neuromuscular blockade in all patients.
* Maintenance of general anesthesia: balanced anesthesia will be administered for maintenance at the anesthesiologists' discretion. We suggest the following regimen: sevoflurane (0.5-1 MAC), remifentanil IV 0.05-0.25 μg/kg/min, and propofol IV 20-75 μg/kg/min. In accordance with guidelines for Good Clinical Practices in pharmacodynamic studies of NMBA, neuromuscular monitoring will be assessed via the train-of-four (TOF) stimulation. TOF device will be placed on the ulnar nerve to illicit twitches in the adductor pollicis. The response to TOF stimulation will be assessed by the anesthesiologist every 30 minutes, starting at intubation. If second response reappears in the TOF stimulation, supplemental doses of rocuronium will be administered at anesthesiologists' discretion.
* Neuromuscular blockade reversal: after peritoneal (port sites) closure, TOF will be assessed. Exact doses of the study medications (previously determined by total body weight) will be administered as following:

  * Sugammadex:

    * If spontaneous recovery has reached second twitch after TOF: 2 mg/kg
    * If spontaneous recovery has reached between 1-2 post-tetanic counts but no twitch responses to TOF: 4 mg/kg
    * When there is a clinical need to reverse NMB within 3 min of a single dose of rocuronium (1.2 mg/kg): 16 mg/kg
  * Neostigmine: 50 µg. Kg-1 will be administered after spontaneous recovery has reached fourth twitch after TOF in accordance with our institutional standard procedures and published literature [10, 11]
* After IP administration, TOF will be assessed every 30 seconds during the first 3 minutes and every minute afterwards to TOF value ≥ 0.9
* The following variables will be collected:

  * Time from peritoneal closure (port sites) to anesthesia readiness for OR discharge to PACU
  * Time from IP administration to extubation
  * Time from IP administration to TOF ≥ 0.9
  * Time from IP administration to anesthesia readiness for OR discharge to PACU II.4.C. Postoperative phase (Postoperative Care Unit)
* The modified Aldrete score will be documented in the EMR.
* Time to discharge-readiness from the OR to PACU, admission time to PACU, and time to discharge from the hospital will be recorded.
* Perioperative incidence of IP related adverse events (i.e. bradycardia, anaphylaxis, nausea and vomiting, and hypotension) Summary statistics will be calculated and reported as means (standard deviations) or medians [inter-quartile ranges] for continuous variables and as frequencies (percentages) for categorical variables. Study groups will be compared using Student's t-tests or Wilcoxon Rank-Sum tests for continuous variables and chi-squared or Fisher's exact tests for categorical variables where appropriate. Primary hypotheses comparing time from peritoneal closure (port sites) to anesthesia readiness for OR discharge to PACU between study groups will be tested using Student's unpaired t-tests (on the natural log transformed outcomes if necessary) at the 5% type I error rate. All analyses will be conducted using SAS version 9.4 (SAS Institute, Cary, N.C.) The study will last approximately one year including recruitment, analysis of the data and writing of the manuscript.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects undergoing outpatient surgeries (laparoscopic cholecystectomy, laparoscopic hernia repair, laparoscopic appendectomy) under general anesthesia requiring rocuronium-induced neuromuscular blockade
2. Male or female patient 18 years and older
3. Able to consent
4. American Society of Anesthesiologist (ASA) physical status of I, II, or III

Exclusion Criteria:

1. Participating in another interventional study drug within 30 days prior to their recruitment
2. Special population (Pregnant, Inmate, Breastfeeding)
3. History of allergy to sugammadex or rocuronium
4. Any medication known to interfere with NMBA or sugammadex
5. Presence of any clinical condition as determined by the investigator that exclude the patient from the trial such as COPD, CKD, and neuromuscular or neurodegenerative diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Sugammadex blockade reversal reduce discharge to PACU. | 1 hour
  Time from peritoneal closure (port sites) to anesthesia readiness for OR discharge to PACU

SECONDARY OUTCOMES:
Extubation time | 1 hour
  Time from IP administration to extubation
TOF less than 0.9 | 1 hour
  Time from IP administration to TOF ≥ 0.9
PACU | 1 hour
  Time from IP administration to anesthesia readiness for OR discharge to PACU

CONTACTS AND LOCATIONS:
Overall Officials: Sergio D Bergese, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sokol-Kobielska E. Sugammadex - indications and clinical use. Anaesthesiol Intensive Ther. 2013 Apr-Jun;45(2):106-10. doi: 10.5603/AIT.2013.0023. PMID 23877905
- [Background] Ali HH, Utting JE, Gray C. Stimulus frequency in the detection of neuromuscular block in humans. Br J Anaesth. 1970 Nov;42(11):967-78. doi: 10.1093/bja/42.11.967. No abstract available. PMID 5488360
- [Background] Sundman E, Witt H, Olsson R, Ekberg O, Kuylenstierna R, Eriksson LI. The incidence and mechanisms of pharyngeal and upper esophageal dysfunction in partially paralyzed humans: pharyngeal videoradiography and simultaneous manometry after atracurium. Anesthesiology. 2000 Apr;92(4):977-84. doi: 10.1097/00000542-200004000-00014. PMID 10754616
- [Background] Keating GM. Sugammadex: A Review of Neuromuscular Blockade Reversal. Drugs. 2016 Jul;76(10):1041-52. doi: 10.1007/s40265-016-0604-1. PMID 27324403
- [Background] Nag K, Singh DR, Shetti AN, Kumar H, Sivashanmugam T, Parthasarathy S. Sugammadex: A revolutionary drug in neuromuscular pharmacology. Anesth Essays Res. 2013 Sep-Dec;7(3):302-6. doi: 10.4103/0259-1162.123211. PMID 25885973
- [Background] Co, M. Bridion® (sugammadex) injection, for intravenous use: US prescribing information. 2015. 2015 [cited 2016 10 OCT ]; http://www.accessdata.fda.gov/. ].
- [Background] Grintescu, I., et al., Comparison of the cost-effectiveness of sugammadex and neostigmine during general anaesthesia for laparoscopic cholecystectomy. BJA: The British Journal of Anaesthesia, 2009. 103(6).
- [Background] Carron M, Zarantonello F, Tellaroli P, Ori C. Efficacy and safety of sugammadex compared to neostigmine for reversal of neuromuscular blockade: a meta-analysis of randomized controlled trials. J Clin Anesth. 2016 Dec;35:1-12. doi: 10.1016/j.jclinane.2016.06.018. Epub 2016 Aug 4. PMID 27871504
- [Background] Paton F, Paulden M, Chambers D, Heirs M, Duffy S, Hunter JM, Sculpher M, Woolacott N. Sugammadex compared with neostigmine/glycopyrrolate for routine reversal of neuromuscular block: a systematic review and economic evaluation. Br J Anaesth. 2010 Nov;105(5):558-67. doi: 10.1093/bja/aeq269. Epub 2010 Oct 8. PMID 20935005
- [Background] Donati F. Residual paralysis: a real problem or did we invent a new disease? Can J Anaesth. 2013 Jul;60(7):714-29. doi: 10.1007/s12630-013-9932-8. Epub 2013 Apr 27. PMID 23625545
- [Background] Hunter JM. Reversal of residual neuromuscular block: complications associated with perioperative management of muscle relaxation. Br J Anaesth. 2017 Dec 1;119(suppl_1):i53-i62. doi: 10.1093/bja/aex318. PMID 29161387
- [Derived] Fiorda Diaz J, Echeverria-Villalobos M, Esparza Gutierrez A, Dada O, Stoicea N, Ackermann W, Abdel-Rasoul M, Heard J, Uribe A, Bergese SD. Sugammadex versus neostigmine for neuromuscular blockade reversal in outpatient surgeries: A randomized controlled trial to evaluate efficacy and associated healthcare cost in an academic center. Front Med (Lausanne). 2022 Dec 8;9:1072711. doi: 10.3389/fmed.2022.1072711. eCollection 2022. PMID 36569123